CLINICAL TRIAL: NCT06333990
Title: A Randomized Clinical Trial of Quetiapine to Reduce Post Concussive Syndrome Polypharmacy
Brief Title: Quetiapine to Reduce Post Concussive Syndrome After Mild Traumatic Brain Injury (mTBI)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Foundation for Advancing Veterans' Health Research (Other)
Collaborators: The University of Texas Health Science Center at San Antonio (Other); Biomedical Research Institute of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20220796HU
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Mild Traumatic Brain Injury
Keywords: Post Concussive Syndrome (PCS); Posttraumatic Stress Disorder (PTSD); Polypharmacy; Quetiapine; Veterans
MeSH Terms: conditions — Brain Concussion; Post-Concussion Syndrome; Stress Disorders, Post-Traumatic | interventions — Quetiapine Fumarate; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Quetiapine (Experimental): Quetiapine will be cross-tapered up to a maximum dose of 200 mg (as tolerated) as other standard of care medications are discontinued.
  Interventions: Drug: Quetiapine Fumarate
- Treatment As Usual (TAU) (Active Comparator): Participants in the TAU group will have doses adjusted over the same period as indicated by usual care criteria.
  Interventions: Drug: TAU

INTERVENTIONS:
Drug: Quetiapine Fumarate — Quetiapine is an atypical antipsychotic approved by the FDA for the treatment of schizophrenia, bipolar disorder, and as an adjunct to treat major depression. It has a broad spectrum of actions at dopaminergic (D1, D2, D3 and D4), serotonergic (5-HT2A, 5-HT2C and 5-HT7), adrenergic (α1), histaminic (H1) and muscarinic (mACh), and partial agonist at 5-HT1A receptors.
  Other Names: Seroquel
  Arms: Quetiapine
Drug: TAU — Standard of care psychotropic medications for treatment of patients with mTBI.
  Other Names: Treatment As Usual
  Arms: Treatment As Usual (TAU)

SUMMARY:
A two site, 2-arm, Phase III randomized pragmatic clinical trial evaluating the effectiveness of quetiapine monotherapy in comparison to Treatment As Usual (TAU) medication management for symptoms experienced by veterans receiving rehabilitation therapy for mild traumatic brain injury (mTBI) and comorbid symptoms of posttraumatic stress disorder (PTSD).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female veterans seeking treatment for mTBI, aged 18-65 years
2. Meet mTBI diagnosis and have PCS symptoms reported on the Neurobehavioral Symptom Inventory (NSI). Six months or more must elapse between the injury and Screening. mTBI diagnosis will be determined using the provisional diagnostic convention recommended by the VA/DoD requiring loss of consciousness, or a period of altered consciousness, or posttraumatic amnesia;
3. Be stable (i.e., no dose changes for > 1 month) on at least three CNS active psychotropic medications prescribed for symptom relief or psychiatric treatment.
4. Have posttraumatic symptoms measured by PTSD Checklist for DSM-5 (PCL-5) score ≥25.

Exclusion Criteria:

1. Moderate or severe TBI, or major neurocognitive disorder (dementia).
2. Meet DSM-5 criteria for schizophrenia, bipolar disorder, schizoaffective disorder, or requiring inpatient hospitalization currently or within past 6 months.
3. Currently taking any antipsychotics or prohibited medication within the past month .
4. Known intolerance to quetiapine or a history of clinically unstable heart, lung, liver, renal, hematological, or endocrinological condition, diabetes mellitus, severe sleep apnea and/or seizure disorder.
5. Substance use disorder severe enough to require medication treatment or medical detoxification or inpatient hospitalization within 6 months of screening.
6. Reporting suicidal ideation of type 4 or 5 in the Columbia Suicide Severity Rating Scale (CSSRS) in the past 3 months prior to screening or at screening or baseline visit (i.e. active suicidal thought with method and intent but without specific plan, or active suicidal thought with method, intent, and plan); or homicidal ideation with intent or plan to harm others within 90 days or suicide attempt; or suicidal behavior within 6 months prior to screening.

   (Note: Study psychiatrist will be immediately notified when SI or HI intent is positive)
7. Current or known history of cardiac arrhythmia or QTc interval ≥ 470 milliseconds.
8. Pregnant or lactating women and those of child-bearing potential not using a reliable method of contraception will be excluded from participating in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Neurobehavioral Symptom Inventory | 2 weeks
  A 22- item, self-report measure of symptoms of postconcussive symptoms severity for the preceding 2 week period. Items are scored on a 5-point scale, and a total score is obtained by summing the 22 symptom items, with higher scores indicate greater symptom severity. The total scores range from 0 - 88.
World Health Organization Disability Assessment Scale | 30 days
  A 12-item, self-report measure of functional disability for the preceding 30 days. Items are scored on a 5-point scale, and a total score is obtained by summing the 12 activities, with higher scores indicate greater disability. The total scores range from 0 - 48.
World Health Organization Quality of Life BREF | 2 weeks
  A 26- item, self-report measure to assess functioning and quality of life for the preceding 2 week period. It is a measure of conceptual domains of quality of life: material and physical well-being, relationships with other people, social, community and civic activities, personal development and fulfillment, independence, and recreation.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - New Mexico VA Healthcare System, Albuquerque, New Mexico
  - South Texas Veterans Healthcare System, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
All de-identified IPD will be shared with the research community through Federal Interagency Traumatic Brain Injury Research (FITBIR) Informatics System.
Supporting Information: SAP
Time Frame: Anticipated June 2028